CLINICAL TRIAL: NCT00452036
Title: Prospective Study to Find a Diagnostic Algorithm for Diagnosis of Minor Head Injury
Brief Title: Diagnostic Algorithm in Patients With Minor Head Injury
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Harald Wolf, Department for Trauma Surgery
Other Study IDs: HW2
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Minor Head Injury; Traumatic Brain Injury
Keywords: risk factors; plain x ray; cranial computed tomography; minor head injury
MeSH Terms: conditions — Craniocerebral Trauma; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Minor head injury: patients with minor head injury
- minor head injury: patients with minor head injury

SUMMARY:
The objective of this prospective study is to evaluate the reliability of plain x-rays vs.cranial computed tomography as a screening method for skull fractures and its prognostic value for intracranial bleeding (ICB).

DETAILED DESCRIPTION:
In a consecutive patients series of about 12500, blunt head injuries were observed (during a 16 month period), in a prospective analysis.

Based on a retrospective study, we created a checklist of individual patients data which was completed for each patient.

In accordance with the institutions guidelines all patients with blunt head injury received plain skull x-ray in 2 plains and additional cranial CT-scan (CCT) in case of fracture or neurological symptoms. We developed also an diagnostic algorithm consisting of anamnestical data and clinical signs and symptoms to define these risk factors and to catch all patients with minor head injury who are at risk to develop intracranial bleeding.

ELIGIBILITY:
Inclusion Criteria:

* head injury, nausea, vomiting

Exclusion Criteria:

* no head injury

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients seen in the trauma outpatient area
Sampling Method: Non-Probability Sample
Enrollment: 12500 (Actual)
Dates: Start 2004-12; Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harald C. Wolf, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Department for Traumatology/Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Stiell IG, Lesiuk H, Wells GA, McKnight RD, Brison R, Clement C, Eisenhauer MA, Greenberg GH, MacPhail I, Reardon M, Worthington J, Verbeek R, Rowe B, Cass D, Dreyer J, Holroyd B, Morrison L, Schull M, Laupacis A; Canadian CT Head and C-Spine Study Group. The Canadian CT Head Rule Study for patients with minor head injury: rationale, objectives, and methodology for phase I (derivation). Ann Emerg Med. 2001 Aug;38(2):160-9. doi: 10.1067/mem.2001.116796. PMID 11468612
- [Background] Stiell IG, Lesiuk H, Wells GA, Coyle D, McKnight RD, Brison R, Clement C, Eisenhauer MA, Greenberg GH, Macphail I, Reardon M, Worthington J, Verbeek R, Rowe B, Cass D, Dreyer J, Holroyd B, Morrison L, Schull M, Laupacis A; Canadian CT Head and C-Spine Study Group. Canadian CT head rule study for patients with minor head injury: methodology for phase II (validation and economic analysis). Ann Emerg Med. 2001 Sep;38(3):317-22. doi: 10.1067/mem.2001.116795. PMID 11524653
- [Background] Stiell IG, Wells GA, Vandemheen KL, Clement CM, Lesiuk H, De Maio VJ, Laupacis A, Schull M, McKnight RD, Verbeek R, Brison R, Cass D, Dreyer J, Eisenhauer MA, Greenberg GH, MacPhail I, Morrison L, Reardon M, Worthington J. The Canadian C-spine rule for radiography in alert and stable trauma patients. JAMA. 2001 Oct 17;286(15):1841-8. doi: 10.1001/jama.286.15.1841. PMID 11597285
- [Background] Haydel MJ, Preston CA, Mills TJ, Luber S, Blaudeau E, DeBlieux PM. Indications for computed tomography in patients with minor head injury. N Engl J Med. 2000 Jul 13;343(2):100-5. doi: 10.1056/NEJM200007133430204. PMID 10891517
- [Background] Miller EC, Holmes JF, Derlet RW. Utilizing clinical factors to reduce head CT scan ordering for minor head trauma patients. J Emerg Med. 1997 Jul-Aug;15(4):453-7. doi: 10.1016/s0736-4679(97)00071-1. PMID 9279694